CLINICAL TRIAL: NCT02929771
Title: Using Virtual Reality to Reduce Procedural Pain in Children With Cancer: A Pilot Randomized Controlled Trial
Brief Title: Using Virtual Reality to Reduce Procedural Pain in Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jennifer Stinson, Clinician Scientist, Clinical Nurse Specialist/NP, PhD, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1000053757
Record Dates: First submitted 2016-10-07; First posted 2016-10-11 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Cancer
Keywords: Virtual Reality; Subcutaneous Port Sampling; Pain; Children
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In addition to usual care, the intervention group will receive the Samsung GearVR with head mounted display (HMD), controller, and headphones. They will situated in front of the nurse and beside/on the lap of the parent, or they may be lying supine. The VR intervention will use auditory and visual stimuli (simulating the peaceful underwater environment) to distract the child before, during, and after the SCP needle insertion. Children will be allowed to 'try-out' the VR system before the SCP access to familiarize themselves with the equipment. The entire study will be videotaped.
  Interventions: Device: Samsung GearVR
- Control Group (Active Comparator): In addition to usual care, participants in the control group will be seated with their parent and in front of the nurse, according to preference. Children will watch an age appropriate video selected by an oncology-affiliated child life specialist on an iPad, while wearing the same headphones used in the experimental condition. The RA will hold the iPad and positioned within a meter of the child so that the child can still see the iPad without the RA interfering in the clinical procedure. The entire study will be videotaped.
  Interventions: Device: iPad

INTERVENTIONS:
Device: Samsung GearVR — VR with head mounted display (HMD) and headphones. Treatment
  Arms: Intervention Group
Device: iPad — iPad with headphones. Control
  Arms: Control Group

SUMMARY:
This study will assess the impact of virtual reality (VR) in decreasing procedural pain related to subcutaneous port (SCP) access in children with cancer. The study is a pilot-randomized controlled trial (RCT) using a cross-over design that will provide us with detailed information on the feasibility of implementing our trial protocol in a future multi-center RCT as well as preliminary estimate of VR treatment effect on children with cancer undergoing SCP access, including child and parent factors potentially associated with VR distraction treatment efficacy.

DETAILED DESCRIPTION:
The study is a repeated-measures cross-over pilot RCT to examine the feasibility of the trial protocol for a study into the effectiveness of immersive VR in minimizing procedural pain and distress in children with cancer. The research objectives are to: (1) pilot implementing immersive virtual reality (VR) for effectiveness testing in a future RCT (measured as implementation outcomes); (2) determine treatment effect sizes (measured as preliminary effectiveness outcomes), between VR, programmed to distract children during an SCP needle insertion, and an active control intervention (i.e., watching a video with headphones); and (3) assess impact of child and parent factors potentially associated with VR treatment effectiveness. Both the intervention and control groups will receive standard medical care (e.g., topical anesthetics). A convenience sample of 40 children and adolescents with cancer (20 participants per treatment arm; 10 boys and 10 girls per treatment arm) will be recruited. In addition, each child will act as their own control. A washout period of 1 month will be used to control for any carry-over effect between conditions. In addition to usual care, children in the experimental condition will wear the VR headset plus headphones. In the control condition, children will watch a video (i.e., an age-appropriate video selected by an oncology-affiliated child life specialist) on an iPad, while wearing the same headphones as in the experimental condition. Implementation outcomes include accrual and retention rates, acceptability and technical difficulties. Effectiveness outcomes include child pain, distress, and fear, as well as parent distress.

ELIGIBILITY:
Inclusion Criteria:

* Child and parent able to speak and understand English
* actively undergoing cancer treatment
* being less than 1 year from initial diagnosis
* requiring at least 2 SCP needle insertions for cancer treatment over the following 8 weeks

Exclusion Criteria:

* visual, auditory or cognitive impairments precluding interaction with the intervention or control equipment
* patients with major co-morbid medical or psychiatric conditions (including needle-phobia_ as per their healthcare provider or parent
* end of life patients
* patients with a MRSA infection or symptoms of respiratory or gastrointestinal infection as per any member of their healthcare team which could contaminate the intervention or control equipment
* participation in usability study

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Accural Rates/Retention Rates | 6 months
  Using a recruitment log to measure eligible children per recruitment day, reasons for ineligibility, reasons for non-participation and reasons for study attrition.
Acceptability | 6 months
  Measured using the VR Distraction Satisfaction Questionnaire completed by children and nurses and will collect data on acceptability, perceived utility of pain reducing procedures, and recommendations for changes related to the needle insertion experience.
Outcome measure feasibility | 6 months
  Will be measured as the percentage of completed outcome measures at baseline and study completion and will be recorded on the VR Distraction Activity Log
Technical Difficulties/Practical Difficulties | 6 months
  Record data related to technical/practical difficulties associated with the VR intervention, RA observed difficulties in implementing the trial protocol in the clinic and time to complete SCP access.

SECONDARY OUTCOMES:
Pain Intensity | 6 months
  For both pre and post study procedures, children will self report their pain and parents, nurses and the RA will report children's pain using an 11 point NRS scale (0 being no pain at all and 10 being the most pain you can imagine this child or you having)
Child Distress | 6 months
  For both pre and post study procedures, distress during the SCP study will be measured using the observer-rated Behavioural Approach-Avoidance Scale (BAADS). 2 research team members will code video-recordings from all SCP needle insertion using the BAADS.
Child Fear | 6 months
  Children will report fear both prior to and following the procedure using the CFS which is a visual scale with established psychometrics in children as young as 5.
Child Pain Catastrophizing | 6 months
  Children will report baseline tendencies to catastrophize about pain using the PCS-C.
Parent Pain Catastrophizing | 6 months
  Parents will report baseline tendencies to catastrophize about their child's pain using the PCS-P which is a self-reporting measure of pain.
Parent Distress | 6 months
  Parents will report on their own level of distress following the child's procedure using the Parent Distress Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Stinson, RN, NP, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes